CLINICAL TRIAL: NCT00169026
Title: Alcoholism and Schizophrenia: Effects of Clozapine
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Harvard Medical School (HMS and HSDM) (Other); Commonwealth Research Center, Massachusetts (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Alan Green, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AA11904
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Schizophrenia; Dual Diagnosis; Schizoaffective Disorder; Psychotic Disorder; Substance Abuse; Alcohol Abuse
Keywords: Clozapine; Atypical Antipsychotic; Conventional antipsychotic; Schizophrenia; Dual Diagnosis; Substance Abuse; Alcohol Abuse
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Substance-Related Disorders; Alcoholism | interventions — Congresses as Topic

INTERVENTIONS:
Drug: Clozapine versus typical (conventional) and atypical antipsychotic medications

SUMMARY:
The purpose of this study is to examine the short - term effects of clozapine on alcohol use in persons with schizophrenia and an alcohol use disorder. The hypothesis is that clozapine will have greater efficacy in reducing alcohol use than other antipsychotic medications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* Current diagnosis of an alcohol use disorder with active use in the last 30 days.
* The participant (or the participant's authorized legal representative) understands the nature of the study and has he/she signed an informed consent.
* Ages 19-65.
* Taking olanzapine, risperidone, quetiapine or a typical antipsychotic agent for at least 8 weeks prior to study randomization
* If taking depot medication, at least 3 injection cycles since the last injection prior to study randomization.

Exclusion Criteria:

* Contraindication to clozapine
* Women who are currently pregnant or who desire to become pregnant during the course of the study.
* Current and past treatment with clozapine
* Current treatment with agents proposed to curtail substance use (e.g., disulfiram, naltrexone, acamprosate, buspirone) and agents contraindicated for use with clozapine (e.g., inderal, tegretol, lithium).
* Meets DSM-IV criteria for current dependence of substances other than alcohol.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64
Dates: Start 1999-05; Study Completion 2004-01

PRIMARY OUTCOMES:
Self report using the weekly Time Line Follow Back; Alcohol Use Scale and Drug Use Scale obtained by clinician and key informant; breathalyzer and urine drug screen. Monthly consensus in substance use rating; monthly CDT and clozapine blood levels.

SECONDARY OUTCOMES:
Clinical Measures: Brief Psychiatric Rating Scale; Scale for the Assessment of Negative Symptoms; and Clinical Global Impression; neurological side affects, cognitive assessment and quality of life measure.

CONTACTS AND LOCATIONS:
Overall Officials: Alan I Green, MD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Commonwealth Research Center, Jamaica Plain, Massachusetts, United States

REFERENCES:
- [Background] Green AI, Zimmet SV, Strous RD, Schildkraut JJ. Clozapine for comorbid substance use disorder and schizophrenia: do patients with schizophrenia have a reward-deficiency syndrome that can be ameliorated by clozapine? Harv Rev Psychiatry. 1999 Mar-Apr;6(6):287-96. doi: 10.3109/10673229909017206. PMID 10370435